CLINICAL TRIAL: NCT03718663
Title: Kliniske Smertetests Som prædiktorer for Effekten af GLA:D®-træningsforløb Hos Patienter Med Symptomgivende Slidgigt i knæene
Brief Title: Predictors for Analgesic Effect to Standardized Exercise Therapy for Osteoarthritic Pain
Status: Completed | Type: Observational
Sponsor: Kristian Kjær Petersen (Other)
Responsible Party: Sponsor-Investigator, Kristian Kjær Petersen, Associated professor, Aalborg University
Organization: Aalborg University (Other)
Other Study IDs: N-20170070
Record Dates: First submitted 2018-10-11; First posted 2018-10-24 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis, Knee; Healthy Subjects
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Knee OA patients (part 1): Painful knee OA patients signed up for standardized exercise therapy
  Interventions: Other: Physiotherapy-guided Evidence-based Exercise Therapy
- Healthy subjects (part 2): Healthy subjects (age 18-28) signed up military service in Defence Command Denmark
  Interventions: Other: Part 2: Military training

INTERVENTIONS:
Other: Physiotherapy-guided Evidence-based Exercise Therapy — Standardized supervised exercise therapy for 6-8 weeks (two times per week).
  Groups: Knee OA patients (part 1)
Other: Part 2: Military training — Part 2: standardized military training for 6-8 weeks in Defence Command Denmark
  Groups: Healthy subjects (part 2)

SUMMARY:
Pain sensitization has been associated with pain severity in people with knee osteoarthritis (KOA) and a neuropathic pain component has been identified in up to 30% of KOA patients. In addition, exercise-induced hypoalgesia (EIH), a measure of descending pain control, has previously been found dysfunctional in a subgroup of people with painful KOA and has also been utilized as a predictive factor for pain progression following total knee replacement.

Measures of pain sensitization have been used prognostic to identify responders to treatment but EIH as a prognostic tool for Physiotherapy-guided Evidence-based Exercise Therapy (PEET) has not been investigated. The primary aim of this explorative study is to investigate if EIH assessed pre-PEET was associated with changes in pain, disability and PainDETECT (PDQ) score post-PEET. The secondary aim is to investigate if PEET changes EIH and PDQ score in patients with painful KOA.

Part 2:

Cross-sectional studies indicate, that daily level of activity influence the effectivity of the EIH mechanims, while pain patients (e.g. KOA patients) can have normal of dysfunctional EIH. It has not been investigated if EIH changes after prolonged exercise in healthy subjects. The aim of this secord part of the study, is to investigate if EIH changes after 6-9 weeks of intensive military training in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* The American College of Rheumatology for clinical knee osteoarthritis (excluding radiological OA assessment)

Exclusion Criteria:

* Known factors to influence pain and pain sensitization.

Part 2:

Inclusion Criteria

* starting as recruits in Defence Command Denmark

Exclusion Criteria:

* Known factors to influence pain and pain sensitization.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 patients with knee osteoarthritis scheduled for PEET.
  Part 2 40 healthy subjects (age 18-28) signed up as recruits in Defence Command Denmark
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 1-2 weeks after last exercise session
  Pain measured on a numerical analog scale from 0 (no pain) to 10 (worst pain imaginable)
Part 2: Exercise-induced hypoalgesia (EIH) | 6-8 weeks into standardized pre-planned military training that continues after the tests
  Change in EIH

CONTACTS AND LOCATIONS:
Overall Officials: Kristian K Petersen, PhD, Principal Investigator — Aalborg University
Locations (1):
- Viby Fysioterapi, Viby J, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided